CLINICAL TRIAL: NCT04483661
Title: Development of Systems and Precision Medicine - Take Mood Disorder as an Example.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B-ER-108-058
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-05

CONDITIONS: Mood Disorders
Keywords: mood disorder, neurocognitive function, metabolic disturbances, microbiota-gut-brain axis, genetic variant, pharmacogenomics
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Precision medicine is to achieve individual optimal health care, given the biological mechanisms, genetic variants, and environmental measurements. Take mood disorder (MD) as an example, we aim to develop systems and precision medicine in Taiwanese population.

MD is a very serious and dysfunctional mental disorder. Since MD patients with treatment have high risk of neurocognitive impairment and metabolic disturbances, the therapeutic strategies are of clinical importance. Individual difference of treatment outcome in MD patients would result from genetic variants, environmental factors, and their interactions. Also, the treatment outcome of MD contains multiple dimensions, including improvement of disease severity, neurocognitive function, and optimized medication strategy. However, comprehensive development of approaches to investigate the multiple dimensions of treatment outcome in MD patients is limited. In this three-year proposal, we explore the interactions of genetic variants and environmental factors (represented by psychosocial stress and gut microbiota) driven approaches to develop precision medicine.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, 20- 70 years of age
* Major depression disorder who met the DSM-V diagnostic criteria were enrolled
* Subjects take at least one kind of antidepressant.

Exclusion Criteria:

* Pregnant or breast-feeding
* Presence of any other major psychiatric illness
* History of substance and alcohol abuse or dependence
* Presence of auto-immune disorder and infectious diseases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who met the criteria will be successively recruited from the National Cheng Kung University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-11-27 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Depression severity | six months
  Clinician rated score by Structure Interview Guide for the Hamilton Depression Rating Scale (17-item)

SECONDARY OUTCOMES:
The influence of environmental factor in mood disorder | six months
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota
cognitive function assessed using the Finger Tapping Test (FTT) | six months
cognitive function assessed using Wisconsin Card Sorting Test (WCST) | six months
cognitive function assessed using Continuous Performance Test (CPT) | six months

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University (NCKU) Hospital, Tainan, Taiwan